CLINICAL TRIAL: NCT05649852
Title: Anxiolytic Effects of Socio-aesthetics in Cancer Patients Undergoing Chemotherapy (PASITHEA)
Brief Title: Anxiolytic Effects of Socio-aesthetics in Cancer Patients Undergoing Chemotherapy
Acronym: PASITHEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A01822-41
Record Dates: First submitted 2022-11-15; First posted 2022-12-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy Effect
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Other): Adjuvant chemotherapy treatment
  Interventions: Other: Socio-aesthetic care; Other: Supportive care

INTERVENTIONS:
Other: Socio-aesthetic care — Group A (Socio-aesthetic care): 3 sessions carried out by a socio-esthetician, during the first administration of chemotherapy.
Other: Supportive care — Group B (control) will not benefit of socio-aesthetic care during chemotherapy but will benefit all existing support care in the center and accessible to patients: psychology consultation, sophrology, art therapy, physiotherapy, hypnosis. The patient will receive support care (maximum 2) during the intercure.

SUMMARY:
The purpose of the study is to assess the average of the "State Anxiety" score of the State Trait Inventory Anxiety at the end of the third cycle of chemotherapy compared to the pre-treatment score (inclusion)

DETAILED DESCRIPTION:
As part of this study, patients will be seen 6 times for the purposes of the study: on inclusion, during the first four courses of chemotherapy and at the end of chemotherapy.

The study is offered to the patient during the consultation with the oncologist before the start of chemotherapy. It may possibly be proposed at the latest when he enters hospitalization for chemotherapy.

Two cohorts of patients will be included:

* Patients treated with chemotherapy every 21 days for lung, breast, digestive, colorectal or gynecological cancer;
* Patients treated with chemotherapy every 14 days for digestive or other cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer treated with adjuvant chemotherapy with an interval of 14 or 21 days for the first 3 cycles;
* Chemotherapy naïve patient;
* Patient speaking and understanding French and able to complete the questionnaires;
* Patient having been informed and having signed an informed consent form to participate in the study.

Exclusion Criteria:

* Patient who has already benefited from socio-aesthetic care;
* Protected patient (under legal protection, or deprived of liberty by judicial or administrative decision);
* Patient unable to understand the information related to the study (linguistic, psychological, cognitive reasons, etc.);
* Pregnant or likely to be pregnant (of childbearing age, without effective contraception) or breastfeeding;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient not benefiting from a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of mean of the "State Anxiety" score of the State Trait Inventory Anxiety | Between the inclusion and the end of the third cycle of chemotherapy (maximum cycle of 21 days)
  Change of mean of the "State Anxiety" score of the State Trait Inventory Anxiety at the end of the third cycle of chemotherapy compared to the pre-treatment score (inclusion)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Drôme Ardèche, Valence, France

IPD SHARING:
Plan to Share IPD: No